CLINICAL TRIAL: NCT03034317
Title: Multi-Center, Concurrent-Controlled, On-Label Study of the NeuRx Diaphragm Pacing System (DPS) in Participants With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: NeuRx Diaphram Pacing System (DPS) Use in Amyotrophic Lateral Sclerosis (ALS)
Acronym: PARADIGM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Synapse Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-1000-51
Record Dates: First submitted 2017-01-13; First posted 2017-01-27 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Diaphragm Pacing
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- NeuRx DPS (Active Comparator): Subjects who have initiated noninvasive ventilation (NIV) and receive the NeuRx diaphragm pacing system (DPS).
  Interventions: Device: NeuRx DPS
- No DPS (No Intervention): Subjects who have initiated noninvasive ventilation (NIV) and do not receive the DPS device.

INTERVENTIONS:
Device: NeuRx DPS — Patients who are diagnosed with ALS, have initiated NIV and choose to have the NeuRx DPS implanted.
  Other Names: Diaphragm Pacing System
  Arms: NeuRx DPS

SUMMARY:
The purpose of this research study is to collect more information about the use, safety, and effectiveness of the NeuRx DPS® in ALS patients.

DETAILED DESCRIPTION:
Characterize the safety and benefit of on-label Humanitarian Device Exemption (HDE) use of DPS in patients with ALS who initiated noninvasive ventilation (NIV).

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or older
* Familial or sporadic ALS diagnosed as possible, laboratory-supported probable, probable, or definite according to the World Federation of Neurology El Escorial criteria
* Bilateral phrenic nerve function clinically acceptable as demonstrated by bilateral diaphragm movement with fluoroscopic sniff test or with phrenic nerve conduction studies
* Chronic hypoventilation was documented by at least one of the following:

  * MIP (respiratory muscle strength) less than 60 cmH2O, or
  * Forced Vital Capacity (FVC) less than 50% predicted, or
  * PaCO2 greater than or equal to 45 mmHg, or
  * Nocturnal SaO2 (arterial oxygen saturation) less than or equal to 88% for at least five continuous minutes
* Initiation of non-invasive ventilation at or before time of enrollment
* Suitable surgical candidate to receive diaphragm pacing stimulation
* Negative pregnancy test in female participants of childbearing potential (treatment group)
* Informed consent from patient or designated representative

Exclusion Criteria:

* FVC less than 45% predicted within 10 days prior to surgery.
* Participation in simultaneous therapeutic clinical trial which could affect the safety or benefit outcomes of this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-12 (Actual)

PRIMARY OUTCOMES:
Survival | 24 months
  Compare the survival of patients who initiated noninvasive ventilation (NIV).and who receive DPS to controls without DPS: (1) concurrent controls; (2) historical controls (e.g., Lechtzin and PRO-ACT databases); and (3) virtual controls (Origent).

SECONDARY OUTCOMES:
Relationship between survival time and clinical features of ALS | 24 months
  Determine whether there is a relationship between survival time and ALS onset type.
Relationship between survival time and ALS assessment scores | 24 months
  Determine whether there is a relationship between survival time and Upper Motor Neuron (UMN)/ Lower Motor Neuron (LMN) assessment scores.
Relationship between survival time and onset of weakness from ALS to treatment | 24 months
Relationship between survival time and ALS treatment interventions | 24 months
Relationship between survival time and intraoperative strength of contraction | 24 months
Characterize change in overall and respiratory function | 24 months
  Characterize longitudinal change in overall function (ALSFRS-R) before and after treatment with DPS compared to controls.
Characterize change in respiratory function | 24 months
  Characterize longitudinal change in respiratory function (FVC, MIP) before and after treatment with DPS compared to controls.
Types device and procedure-related adverse events | 24 months
Frequency of device and procedure-related adverse events | 24 months
Types of respiratory serious adverse events | 24 months
Frequency of respiratory adverse events | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Miller, MD, Principal Investigator — California Pacific Medical Center

IPD SHARING:
Plan to Share IPD: No